CLINICAL TRIAL: NCT03254446
Title: A Phase III Randomized, Double Blind, Parallel Group, Placebo Controlled, Multi-centre, Multinational Study to Evaluate Efficacy and Safety of TRC150094 as an Add On to Standard of Care in Improving Cardiovascular Risk in Subjects With Diabetes, Dyslipidemia and Hypertension
Brief Title: Safety and Efficacy Study of TRC150094 to Improve the CV Risk in Subjects With Diabetes, Dyslipidemia and Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT/P015/CMR/16/03_01
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Diabetes; Dyslipidemias; Hypertension
Keywords: Diabetes; Hypertension; Dyslipidemia; Cardiovascular Risk
MeSH Terms: conditions — Diabetes Mellitus; Dyslipidemias; Hypertension | interventions — TRC150094

STUDY DESIGN:
Intervention Model Description: Randomized, Double Blind, Parallel Group, Placebo Controlled, Multi-centre, Multinational Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRC150094 45 mg (Experimental): TRC150094 45 mg Tablet to be administered orally once a day for 50 weeks
  Interventions: Drug: TRC150094
- Placebo (Placebo Comparator): Matching Placebo Tablet to be administered orally once a day for 50 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRC150094 — TRC150094 Tablet 45 mg
  Arms: TRC150094 45 mg
Drug: Placebo — Matching Placebo Tablet
  Arms: Placebo

SUMMARY:
The phase III trial is designed with an aim of determining the efficacy of Investigational Product TRC150094 in concurrently reducing non-traditional risk factors for CV risk i.e., HbA1c, MAP and non-HDL cholesterol. This study will be a randomized, double blind, parallel group, placebo controlled, multi-centre, multinational study in 1250 subjects. All the study subjects will receive once daily dose of TRC150094 45 mg or placebo tablets in addition to their standard of care, for 24 weeks followed by roll over to a safety extension phase of 26 weeks.

DETAILED DESCRIPTION:
TRC150094 is an Investigational Product for the treatment of CV risk associated with non-traditional risk factors ie, diabetes, hypertension and dyslipidemia, which acts by increasing the energy expenditure and restoring mitochondrial flexibility which is deranged in patients with these risk factors. Treatment with TRC150094 has shown clinically meaningful benefits in well-established contributors of CV risk i.e., insulin resistance and hyperglycemia, SBP as well as non-traditional risk factors i.e. non-HDL cholesterol and MAP, over and above standard of care.

The phase III trial is designed with an aim of determining the efficacy of TRC150094 in concurrently reducing non-traditional risk factors for CV risk i.e., HbA1c, MAP and non-HDL cholesterol. This study will be a randomized, double blind, parallel group, placebo controlled, multi-centre, multinational study in 1250 subjects. All the study subjects will receive once daily dose of TRC150094 45 mg or placebo tablets in addition to their standard of care, for 24 weeks followed by roll over to a safety extension phase of 26 weeks.

Primary Objective of the study is, To evaluate the efficacy of TRC150094 in improving cardiovascular (CV) risk in subjects with diabetes, dyslipidemia and hypertension Secondary Objectives of the study are,

1. To evaluate safety of TRC150094 in subjects with diabetes, dyslipidemia and hypertension
2. To evaluate extended safety profile of TRC150094 beyond 24 weeks of treatment in subjects with diabetes, dyslipidemia and hypertension

In this study there will be five visits at week 4, 12, 24, 36 and 50 after enrolment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects in the age range 30-70 years (both inclusive)
2. BMI in the range 23-39 (inclusive) kg/m2
3. HbA1C ≥7.5 %
4. Stable therapy of ≤2 oral hypoglycemic agents for at least two months prior to screening at doses that are appropriate for the duration of the study in the judgment of the investigator.
5. Non HDL-cholesterol ≥ 160 mg/dL.
6. Mean Arterial Pressure (MAP) ≥100 mm Hg based on average of 24 hours' ambulatory blood pressure monitoring (ABPM) with or without antihypertensive treatment (subjects will have to be on stable dose of anti-hypertensive treatment for at least two months prior to screening); Dose should be appropriate for the duration of the study in the judgment of the investigator.
7. Willing to give written informed consent
8. Ability to adhere to the study restrictions and assessments schedule

Exclusion Criteria:

1. Uncontrolled hypertension: SBP of ≥ 180 mm Hg and DBP ≥ 110 mmHg based on average of 24 hours' ambulatory blood pressure monitoring.
2. HbA1C > 10 % at screening.
3. Serum triglycerides >400 mg/dL.
4. LDL-cholesterol >300 mg/dL or medical history/clinical evidence of familial hyperlipidemic disorder.
5. Subjects on Insulin or Sodium Glucose Co-Transporter 2 (SGLT2) inhibitors.
6. Acute coronary syndrome (ACS) or stroke or any revascularization within last 6 months.
7. Subjects having untreated thyroid dysfunction (TSH <0.3 or >5.5 µIU/mL) or hormone related obesity disorder.
8. Subjects with liver enzymes (SGOT, SGPT) more than 3X of upper limit of normal value.
9. eGFR <30 mL/min as evaluated by Modification of Diet in Renal Disease (MDRD) method.
10. Seropositive for HIV, Hepatitis B or Hepatitis C.
11. History of alcohol or drug abuse, psychiatric disorder, any bleeding disorder, malignancy in last 3 years.
12. Pregnant or lactating women.
13. Female of childbearing potential, who are neither surgically sterilized nor willing to use reliable contraceptive methods (double barrier methods or intrauterine device).
14. Male subjects with partners of childbearing potential not willing to use reliable contraception methods.
15. Clinically significant abnormal physical findings, laboratory results, ECG findings and/or any other clinical observation or history during the screening examination, which would interfere with the objectives of the study.
16. Intake of any investigational drug within 3 months prior to the first dose of study drug.
17. In the opinion of the investigator, subject is unable to cooperate with any study procedures, unlikely to adhere to the study procedures, keep appointments, or plan to relocate during the study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Estimated)
Dates: Start 2018-03-12 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change in mean arterial pressure (MAP), non-HDL cholesterol and HbA1c | 24 Weeks
  Mean change in weighted average composite score of change in mean arterial pressure (MAP), non-HDL cholesterol and HbA1c from baseline to 24 weeks of treatment between arms
Change in Joint British Society recommendations on the prevention of cardiovascular disease 3rd iteration (JBS3) risk score | 24 Weeks
  Mean change in Joint British Society recommendations on the prevention of cardiovascular disease 3rd iteration (JBS3) risk score at the end of 24 weeks of treatment between arms

SECONDARY OUTCOMES:
Change in MAP | 24 Weeks
  Mean change in MAP from baseline to 24 weeks of treatment
Change in non-HDL cholesterol | 24 Weeks
  Mean change in non-HDL cholesterol from baseline to 24 weeks of treatment
Change in HbA1c | 24 Weeks
  Mean change in HbA1c from baseline to 24 weeks of treatment

OTHER OUTCOMES:
Change in weight | 24 Weeks
  Mean change in weight from baseline to 24 weeks of treatment
Safety profile of TRC150094 | 50 Weeks
  The safety profile of TRC150094 beyond 24 weeks of treatment shall also be reported

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Tandon, M.D., PhD, Study Chair — All India Institute of Medical Sciences
Locations (21):
- Brazil (5):
  - Comitê de ética em Pesquisa do Hospital Pró Cardíaco, Rio de Janeiro, Botafogo
  - Avenida Angélica, São Paulo, CEP
  - Rua Silva Jardim, São Bernardo do Campo, São Paulo
  - Av. Farroupilha, 8001 Prédio 21, Recepção C, Bairro São José - Canoas/RS, Canoas
  - Rua Coronel Aureliano de Camargo,905, Centro,, Tatuí
- India (12):
  - BAPS Pramukh Swami Hospital,, Surat, Gujarat
  - Bangalore Diabetes Centre, No. 426, 4th Cross, 2nd block, kalyan nagar,, Bangalore, Karnataka
  - Government Medical College, Government Medical College Campus,, Calicut, Kerala
  - Lisie Hospital, Kochi, Kerala
  - Indian Institute of Diabetes, Thiruvananthapuram, Kerala
  - Supe Heart and Diabetes Hospital and Research Centre,, Nashik, Maharashtra
  - Medipoint Hospitals Pvt. Ltd, Pune, Maharashtra
  - Ashirwad Hospital & Research Centre, Ulhasnagar, Maharashtra
  - Dayanand Medical College & Hospital, Ludhiana, Punjab
  - S.R Kalla Memorial Gastro and General Hospital, Jaipur, Rajasthan
  - Diabetes ,Thyroid and Endocrine Centre, Jaipur, Rajasthan
  - Apollo Hospitals, PR No. 3-5-836 to 838, Near Old MLA Quarters,, Hyderabad, Telangana
- Philippines (4):
  - De La Salle Heath Sciences Institute, Dasmariñas, Cavite
  - Angeles University Foundation Medical Center, Angeles City, Pampanga
  - St. Paul's Hospital, General Luna, Saint Iloilo City
  - Davao Doctors Hospital, Davao City

IPD SHARING:
Plan to Share IPD: No